CLINICAL TRIAL: NCT04390165
Title: Olfactory and Gustatory Disturbances as a Clinical Presentation of Coronavirus Disease 2019 (COVID-19) Infection in Malaysia - A Nationwide Multicentre Cross-Sectional Study
Brief Title: Malaysian COVID-19 Anosmia Study (Phase 1) - A Nationwide Multicentre Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Hospital Sultanah Bahiyah (Other Government)
Collaborators: Hospital Tuanku Fauziah, Kangar, Perlis (Unknown); Penang Hospital, Malaysia (Other Government); Hospital Raja Permaisuri Bainun (Other Government); Hospital Sungai Buloh, Selangor (Unknown); Kuala Lumpur General Hospital (Other Government); Hospital Tuanku Jaafar, Seremban, Negeri Sembilan (Unknown); Hospital Melaka, Melaka (Unknown); Hospital Enche Besar Hajjah Khalsom, Kluang, Johor (Unknown); Hospital Raja Perempuan Zainab II, Kota Bahru, Kelantan (Unknown); Hospital Sultanah Nur Zahirah, Kuala Terengganu (Other Government); Hospital Tengku Ampuan Afzan, Kuantan, Pahang (Unknown); Sarawak General Hospital (Other); Hospital Queen Elizabeth, Malaysia (Other Government)
Responsible Party: Principal Investigator, Siti Sabzah bt Mohd Hashim, MD, MS (ORL-HNS), Head of Otorhinolaryngology Service, Ministry of Health, Malaysia & Senior Consultant Otorhinolaryngologist, Hospital Sultanah Bahiyah
Other Study IDs: MCO-001; NMRR-20-934-54803 (Other: National Medical Research Register (NMRR), Malaysia)
Record Dates: First submitted 2020-05-10; First posted 2020-05-15 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV Infection; COVID-19; Anosmia; Dysgeusia
Keywords: Cross-sectional study; Prevalence; Otorhinolaryngology; Infectious Diseases; Anosmia; Dysgeusia; Olfactory Disorders; Taste Disorders; COVID-19; SARS-CoV-2; Coronavirus 2019
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Anosmia; Dysgeusia; Communicable Diseases; Taste Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malaysian COVID-19 Cohort: A cohort of COVID-19 positive patients will be recruited from participating Malaysian Ministry of Health-designated COVID-19 treating hospitals across the country.
  Interventions: Other: Patient-Reported Online Questionnaire on Olfactory & Taste Disturbances

INTERVENTIONS:
Other: Patient-Reported Online Questionnaire on Olfactory & Taste Disturbances — This is an online patient-reported questionnaire that examines the presence or absence of olfactory and taste disturbances, the onset of olfactory and taste disturbances in relation to other COVID-19 symptoms, and the temporal evolution of the severity of olfactory and taste disturbances. The occurrence of ear symptoms in COVID-19 infection will also be evaluated in this questionnaire as a secondary outcome. The questionnaire will also have questions relating to the patient's underlying health conditions, risk factors for COVID-19 infection, and demographics.

SUMMARY:
The Malaysian COVID-19 Anosmia Study is a nationwide multicentre observational study to investigate the prevalence and characteristics of olfactory and gustatory/taste disturbances in COVID-19 infection in Malaysia, and to evaluate the predictive value of screening for these symptoms in COVID-19 infection.

This study consists of two phases: the first phase is a cross-sectional study and the second phase is a case-control study. The cross-sectional study is described here (the case-control study is described in a separate ClinicalTrials.gov record).

DETAILED DESCRIPTION:
The world is currently in the midst of the Coronavirus 2019 (COVID-19) pandemic that is caused by a novel coronavirus, Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). According to published cohort studies on COVID-19 infected patients, the most prevalent symptoms consist of fever, dry cough, dyspnoea, sputum production, myalgia, arthralgia, headache, diarrhoea, and sore throat. Recently, there have been concerns of significant viral transmission through asymptomatic, pre-symptomatic or even mildly symptomatic patients.

There is increasing anecdotal evidence from patients and healthcare professionals highlighting isolated loss of sense of smell (anosmia) and taste disturbances (dysgeusia) as atypical symptoms of COVID-19 infection in otherwise asymptomatic patients. In parallel, expert statements from the British Association of Otorhinolaryngology-Head & Neck Surgery (ENT UK), British Rhinological Society, and the American Association of Otolaryngology-Head & Neck Surgery (AAO-HNS) have suggested that olfactory and taste disturbances could be a clinical feature of COVID-19 infection.

Rapidly emerging evidence from Europe, the United Kingdom and the United States have found olfactory and taste disturbances to be highly prevalent in patients diagnosed with COVID-19. In contrast, there is currently limited evidence from Asia on the prevalence of these symptoms in COVID-19 infection.

The aim of this cross-sectional study is to study the prevalence and characteristics of olfactory and taste disturbance in patients with COVID-19 infection in Malaysia. COVID-19 positive patients will be recruited from participating Malaysian Ministry of Health-designated COVID-19 treating hospitals across the country. Participants will answer an online questionnaire to evaluate and characterise these symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years old
2. Laboratory confirmed COVID-19 infection [Reverse Transcription Polymerase Chain Reaction (RT-PCR)]
3. Patients clinically able to answer the questionnaire

Exclusion Criteria:

1. Patients with olfactory or taste/gustatory disorders before the COVID-19 epidemic
2. Patients without a laboratory-confirmed COVID-19 diagnosis
3. Patients in intensive care unit at the time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are adult patients with laboratory-confirmed COVID-19 infection from participating Malaysian hospital sites in this study, since the arrival of COVID-19 infection in Malaysia (January 2020) until present time.
  These patients comprise those who either currently inpatient or already discharged into the community. For patients already discharged into the community, they will be invited to participate by phone call from the hospital treating team. Once verbal consent has been obtained, they a QR code or internet URL link to the online questionnaire website will be sent to these patients.
Sampling Method: Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of olfactory and taste disturbances in COVID-19 patients | Within 2 weeks preceding the diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked regarding whether they experienced symptoms of olfactory and/or taste disturbances
Prevalence of olfactory disturbances in COVID-19 patients | Within 2 weeks preceding the diagnosis of COVID-19 infection
  Percentage of COVID-19 patients experiencing olfactory disturbances (anosmia or hyposmia)
Prevalence of taste disturbances in COVID-19 patients | Within 2 weeks preceding the diagnosis of COVID-19 infection
  Percentage of COVID-19 patients experiencing taste disturbances

SECONDARY OUTCOMES:
Clinical manifestations of study participants | Within 2 weeks preceding the diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked regarding other symptoms they experienced when they were diagnosed with COVID-19 (e.g. headache, nasal congestion, fever, chills, cough, dyspnoea, gastrointestinal symptoms, eye & ear symptoms)
Other pre-existing health conditions | Prior to diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked regarding their pre-existing health conditions (for example, obesity, diabetes, hypertension, cardiac conditions, previous head trauma, chronic rhinosinusitis, etc.)
Rating of baseline sense of smell & taste in COVID-19 patients prior to diagnosis of their infection | Prior to 2 weeks preceding the diagnosis of COVID-19 infection (Baseline)
  In the patient-reported online questionnaire, subjects will be asked to rate their sense of smell and taste before their diagnosis of COVID-19 infection
Rating of sense of smell & taste in COVID-19 patients at time of diagnosis of their infection | Within 2 weeks preceding the diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked to rate their sense of smell and taste at the time of diagnosis of COVID-19 infection
Rating of sense of smell & taste in COVID-19 patients at time of answering questionnaire survey | Up to 6 months
  In the patient-reported online questionnaire, subjects will be asked to rate their sense of smell and taste at the time of answering questionnaire survey

CONTACTS AND LOCATIONS:
Overall Officials: Siti Sabzah Mohd Hashim, MD MS, Study Chair — Hospital Sultanah Bahiyah
Locations (14):
- Malaysia (14):
  - Hospital Enche' Besar Hajjah Khalsom, Kluang, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Tuanku Jaafar, Seremban, Negeri Sembilan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Tuanku Fauziah, Kangar, Perlis
  - Penang Hospital, George Town, Pulau Pinang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - Kuala Lumpur General Hospital, Kuala Lumpur
  - Hospital Melaka, Malacca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Giacomelli A, Pezzati L, Conti F, Bernacchia D, Siano M, Oreni L, Rusconi S, Gervasoni C, Ridolfo AL, Rizzardini G, Antinori S, Galli M. Self-reported Olfactory and Taste Disorders in Patients With Severe Acute Respiratory Coronavirus 2 Infection: A Cross-sectional Study. Clin Infect Dis. 2020 Jul 28;71(15):889-890. doi: 10.1093/cid/ciaa330. No abstract available. PMID 32215618
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Kaye R, Chang CWD, Kazahaya K, Brereton J, Denneny JC 3rd. COVID-19 Anosmia Reporting Tool: Initial Findings. Otolaryngol Head Neck Surg. 2020 Jul;163(1):132-134. doi: 10.1177/0194599820922992. Epub 2020 Apr 28. PMID 32340555
- [Background] Yan CH, Faraji F, Prajapati DP, Boone CE, DeConde AS. Association of chemosensory dysfunction and COVID-19 in patients presenting with influenza-like symptoms. Int Forum Allergy Rhinol. 2020 Jul;10(7):806-813. doi: 10.1002/alr.22579. Epub 2020 Jun 1. PMID 32279441
- [Background] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008
- [Derived] Lee SH, Yeoh ZX, Sachlin IS, Gazali N, Soelar SA, Foo CY, Low LL, Syed Alwi SB, Tengku Kamalden TMI, Shanmuganathan J, Zaid M, Wong CY, Chua HH, Yusuf S, Muhamad D, Devesahayam PR, Ker HB, Salahuddin Z, Mustafa M, Sawali H, Lee HG, Din S, Misnan NA, Mohamad A, Ismail MN, Periasamy C, Chow TS, Krishnan EK, Leong CL, Lim LPF, Zaidan NZ, Ibrahim MZ, Abd Wahab S, Mohd Hashim SS; Malaysian COVID-19 Anosmia Research Group. Self-reported symptom study of COVID-19 chemosensory dysfunction in Malaysia. Sci Rep. 2022 Feb 8;12(1):2111. doi: 10.1038/s41598-022-06029-6. PMID 35136124
- See also: AAO-HNS: Anosmia, Hyposmia, and Dysgeusia Symptoms of Coronavirus Disease | American Academy of Otolaryngology-Head and Neck Surgery — https://www.entnet.org/content/aao-hns-anosmia-hyposmia-and-dysgeusia-symptoms-coronavirus-disease